CLINICAL TRIAL: NCT03587116
Title: AN OPEN-LABEL, NON-INVESTIGATIONAL PRODUCT, LEAD-IN STUDY TO EVALUATE AT LEAST 6 MONTHS OF PROSPECTIVE EFFICACY AND SAFETY DATA OF FACTOR IX OR FACTOR VIII PROPHYLAXIS REPLACEMENT THERAPY IN THE USUAL CARE SETTING OF MODERATELY SEVERE TO SEVERE ADULT HEMOPHILIA B SUBJECTS (FIX:C≤2%) WHO ARE NEGATIVE FOR nAb TO AAV VECTOR-SPARK100 AND MODERATELY SEVERE TO SEVERE HEMOPHILIA A ADULT SUBJECTS (FVIII:C≤1%) WHO ARE NEGATIVE FOR nAb TO AAV VECTOR SB-525 CAPSID (AAV6), PRIOR TO THE RESPECTIVE THERAPEUTIC PH 3 GENE THERAPY STUDIES (See Detailed Description Section for Official Protocol Title)
Brief Title: A Study to Evaluate Prospective Efficacy and Safety Data of Current FIX Prophylaxis Replacement Therapy in Adult Hemophilia B Subjects (FIX:C≤2%) or Current FVIII Prophylaxis Replacement Therapy in Adult Hemophilia A Subjects (FVIII:C≤1%)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: C0371004; 2017-001271-23 (EudraCT Number)
Record Dates: First submitted 2018-06-29; First posted 2018-07-16 (Actual); Results first posted 2025-11-06 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-10

CONDITIONS: Hemophilia B; Hemophilia A
MeSH Terms: conditions — Hemophilia B; Hemophilia A

STUDY DESIGN:
Intervention Model Description: The data obtained from this lead-in study will serve as the control group for the subsequent Phase 3 gene therapy study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Standard of Care FIX replacement therapy (Other)
  Interventions: Drug: Standard of Care FIX Replacement therapy
- Standard of Care FVIII replacement therapy (Other)
  Interventions: Drug: Standard of Care FVIII Replacement therapy

INTERVENTIONS:
Drug: Standard of Care FIX Replacement therapy — There is no investigational product being administered. Subjects will be administering their own standard of care FIX replacement therapy.
  Arms: Standard of Care FIX replacement therapy
Drug: Standard of Care FVIII Replacement therapy — There is no investigational product being administered. Subjects will be administering their own standard of care FVIII replacement therapy.
  Arms: Standard of Care FVIII replacement therapy

SUMMARY:
To establish baseline prospective efficacy data of current FIX prophylaxis replacement therapy in the usual care setting of hemophilia B subjects, who are negative for nAb to AAV-Spark100, prior to the Phase 3 gene therapy study.

To establish baseline prospective efficacy data of current FVIII prophylaxis replacement therapy in the usual care setting of hemophilia A subjects, who are negative for nAb to AAV6, prior to the Phase 3 gene therapy study.

The enrollment for hemophilia A participants is completed. At this time participants are only being enrolled for hemophilia B cohort.

DETAILED DESCRIPTION:
AN OPEN-LABEL, NON-INVESTIGATIONAL PRODUCT, MULTI-CENTER, LEAD-IN STUDY TO EVALUATE PROSPECTIVE EFFICACY AND SELECTED SAFETY DATA OF CURRENT FACTOR IX (FIX) OR FACTOR VIII (FVIII) PROPHYLAXIS REPLACEMENT THERAPY IN THE USUAL CARE SETTING OF MODERATELY SEVERE TO SEVERE ADULT HEMOPHILIA B SUBJECTS (FIX:C≤2%) WHO ARE NEGATIVE FOR NEUTRALIZING ANTIBODIES TO ADENO-ASSOCIATED VIRUS VECTOR-SPARK100 (BENEGENE-1) AND MODERATELY SEVERE TO SEVERE HEMOPHILIA A ADULT SUBJECTS (FVIII:C≤1%) WHO ARE NEGATIVE FOR NEUTRALIZING ANTIBODIES TO ADENO-ASSOCIATED VIRUS VECTOR 6 (AAV6), PRIOR TO THE RESPECTIVE THERAPEUTIC PHASE 3 GENE THERAPY STUDIES

ELIGIBILITY:
Inclusion Criteria:

Hemophilia B Population:

1. Evidence of a signed and dated informed consent document indicating that the participant has been informed of all pertinent aspects of the study.
2. Willing and able to comply with scheduled visits, FIX prophylaxis treatment plan, laboratory tests and other study procedures.
3. Males ≥ 18 and <65 years of age with moderately severe to severe hemophilia B and documented FIX activity (≤2%) prior to baseline visit.
4. Previous experience with FIX therapy (≥50 documented exposure days to a FIX protein product such as recombinant, plasma-derived or extended half-life FIX product).
5. Participants on FIX prophylaxis replacement therapy (recombinant, plasma-derived or extended half-life FIX product) must have the intention to remain on FIX prophylaxis replacement therapy for the duration of the study.
6. No known hypersensitivity to FIX replacement product.
7. No history of FIX inhibitor (clinical or laboratory-based assessment) defined as a titer

   * 0.6 BU/mL, regardless of the laboratory normal range, or any measured Bethesda inhibitor titer greater than the upper limit of normal for the laboratory performing the assay. Clinically, no signs or symptoms of decreased response to FIX administration. Participants will not be required to undergo diagnostic evaluation of inhibitor status to participate in the study.

Hemophilia A Population:

1. Evidence of a signed and dated informed consent document indicating that the participant has been informed of all pertinent aspects of the study.
2. Willing and able to comply with scheduled visits, FVIII prophylaxis treatment plan, laboratory tests and other study procedures.
3. Males ≥18 and <65 years of age with moderately severe to severe hemophilia A and documented FVIII activity (≤1%) prior to baseline visit.
4. Previous experience with FVIII therapy (≥150 documented exposure days to a FVIII protein product such as recombinant, plasma-derived or extended half-life FVIII product).
5. Participants must be on a stable FVIII prophylaxis replacement therapy (recombinant, plasma-derived or extended half-life FVIII product) at study entry and must have the intention to remain on FVIII prophylaxis replacement therapy for the duration of the study. This does not include nonfactor treatments, which are prohibited.
6. No known hypersensitivity to FVIII replacement product.
7. No history of FVIII inhibitor (clinical or laboratory-based assessment) defined as a titer ≥0.6 BU/mL, regardless of the laboratory normal range, or any measured Bethesda inhibitor titer greater than the upper limit of normal for the laboratory performing the assay. Clinically, no signs or symptoms of decreased response to FVIII administration. Participants will not be required to undergo diagnostic evaluation of inhibitor status to participate in the study.

Exclusion Criteria:

1. Anti-AAV-Spark100 neutralizing antibody titer above the established threshold performed by a central laboratory during screening in hemophilia B subjects or Anti-AAV6 neutralizing antibody titer above the established threshold performed by a central laboratory during screening in hemophilia A subjects.
2. Lack of participant compliance with documentation of bleeds and/or prophylaxis replacement therapy administration.
3. If there is no documentation regarding hepatitis status, as defined below, within the last 12 months prior to screening for hepatitis B and 6 months prior to screening for hepatitis C, then participants will be required to have the following hepatitis testing performed at screening:

   1. Hepatitis B screening (acute and chronic):

      HBsAg (also referred to as Hepatitis B surface antigen), HBV-DNA viral assay (also referred to as a nucleic acid test for Hepatitis B virus DNA), and Anti-HBc (also referred to as Total Hepatitis B core antibody).
      * A participant is not eligible if either HbsAg is positive or HBV-DNA is positive/detectable.
      * Anti-HBc must be obtained in all participants for determination of whether the participant had prior hepatitis B. If the anti-HBc is positive and both HBsAg and HBV DNA are negative this would be consistent with a prior infection and the subject would be eligible for the study. Anti-HBc must be obtained in all subjects to discriminate between those with no prior hepatitis B and those with prior infection in the event of reactivation. FDA has noted reactivation of hepatitis B virus exists.
      * One documented negative HBV-DNA viral load is sufficient to assess eligibility. A participant who is currently undergoing anti-viral therapy for hepatitis B is not eligible.
   2. Hepatitis C (acute or chronic):

      * A participant who is currently undergoing anti-viral therapy for chronic hepatitis C is not eligible.
      * Participants treated with anti-viral therapy for chronic hepatitis C, must have completed anti-viral therapy at least 6 months prior to screening and have a negative HCV-RNA at least 6 months prior to screening.
      * All participants (who are not currently undergoing anti-viral therapy for chronic hepatitis C) must have a single HCV-RNA load assay (also referred to as a nucleic acid test [NAT] for HCV RNA) obtained during the 6 months preceding screening. This includes participants with prior known chronic hepatitis C who have completed treatment with anti-viral therapy.
      * A participant is not eligible if his HCV-RNA load assay result is positive/detectable.
4. Currently on antiviral therapy for hepatitis B or C.
5. Significant liver disease, as defined by pre-existing diagnosis of portal hypertension, splenomegaly, or hepatic encephalopathy.

   All participants who do not have the listed pre existing diagnoses above must have the following assessments performed within the last 12 months prior to screening and if not will need to be tested for liver fibrosis status at screening: a serum albumin level below normal limits and/or significant liver fibrosis by any of the following diagnostic modalities: FibroScan median stiffness score >8 kPa units OR FibroTest/FibroSURE >0.48*.

   * NOTE: If there is concern regarding the validity of any of the liver fibrosis test results please contact the medical monitor to discuss whether any additional testing needs to be performed (ie, either repeating any test or performing another fibrosis test). Also, note, if a participant has a known history of Gilbert's syndrome, a FibroTest cannot be used for fibrosis testing.
6. Documented serological evidence of human immunodeficiency virus HIV-1 or HIV-2 with Cluster of Differentiation 4 positive (CD4+) cell count ≤200 mm3 within the last 12 months prior to screening. Participants who are HIV positive and stable, have an adequate CD4 count (>200/mm3) and undetectable viral load (<50 gc/mL) documented within the preceding 12 months, and are on an antiretroviral drug regimen are eligible to enroll. Participants who have not been tested within the prior 12 months of screening will need to be tested for HIV status at screening.
7. History of chronic infection or other chronic disease that the investigator deems an unacceptable risk. In addition, any participant with conditions associated with increased thromboembolic risk such as known inherited or acquired thrombophilia, or a history of thrombotic events including but not limited to stroke, myocardial infarction, and/or venous thromboembolism, is excluded.
8. Any concurrent clinically significant major disease or condition that the investigator deems unsuitable for participation or other acute or chronic medical or psychiatric condition including recent (within the past year) or active suicidal ideation or behavior or laboratory abnormality that may increase the risk associated with study participation or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the participant inappropriate for entry into this study. In addition, any participant with a history of a neoplasm (including hepatic malignancy) that required treatment (eg, chemotherapy, radiotherapy, immunotherapy), is excluded, except for adequately treated basal or squamous cell carcinoma of the skin or a surgically removed benign neoplasm not requiring chemotherapy, radiotherapy and/or immunotherapy. Any other neoplasm that has been cured by resection should be discussed between the investigator and sponsor.
9. Participation in other studies if involving administration of investigational product(s) within the last 3 months prior to study entry and/or during study participation or in a previous gene therapy clinical study within the last 12 months prior to screening.

   • Participants already enrolled in this lead-in study (C0371004) may be allowed to participate in the screening and baseline periods of either C0371002 or C3731003 protocols prior to their completion of the end of study visit in this lead-in study.
10. Any participant who previously received fidanacogene elaparvovec (hemophilia B) or giroctocogene fitelparvovec (hemophilia A) or any AAV gene-based therapy.
11. Participants using restricted therapies.
12. Any participant with a planned surgical procedure requiring FIX (hemophilia B) or FVIII (hemophilia A) surgical prophylactic factor treatment in the next 24 months.
13. Investigator site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, or participants who are Pfizer employees, including their family members, directly involved in the conduct of the study.

NOTE: The sponsor's medical team should be contacted if there are any questions regarding any of the inclusion or exclusion criteria (Sections: 4.1 and 4.2).

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 212 (Actual)
Dates: Start 2018-07-26 (Actual); Primary Completion 2024-12-13 (Actual); Study Completion 2024-12-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (75):
- United States (13):
  - Clinical and Translational Research Unit (CTRU), Palo Alto, California
  - Lucile Packard Childrens Hospital, Palo Alto, California
  - University of California, San Francisco - Outpatient Hematology Clinic, San Francisco, California
  - Stanford Health Care, Stanford, California
  - Hemophilia and Thrombosis Center at the University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Investigational Drug Service, Atlanta, Georgia
  - Indiana Hemophilia & Thrombosis Center, Inc., Indianapolis, Indiana
  - Mississippi Center for Advanced Medicine, Madison, Mississippi
  - Alliance for Childhood Diseases, Las Vegas, Nevada
  - Penn Blood Disorder Center, Philadelphia, Pennsylvania
  - Bloodworks NW, Seattle, Washington
- Australia (5):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - The Alfred Hospital, Melbourne, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
- Cliniques universitaires Saint-Luc/Unité d'Hématology et Hémostase, Brussels, Belgium
- Brazil (6):
  - Centro Estadual de Hemoterapia e Hematologia Marcos Daniel Santos - Hemoes, Vitória, Espírito Santo
  - Centro de Hemoterapia e Hematologia do Para - Fundação HEMOPA, Belém, Pará
  - Centro de Hematologia e Hemoterapia - Hemocentro de Campinas - UNICAMP, Campinas, São Paulo
  - Hospital Das Clínicas Da Faculdade de Medicina de Ribeirao Preto Da Universidade de Sao Paulo, Ribeirão Preto, São Paulo
  - lnstituto Estadual de Hematologia Arthur de Siqueira Cavalcanti - HEMORIO, Rio de Janeiro
  - Hospital das Clinicas da Faculdade de Medicina da Universidade de Sao Paulo, São Paulo
- Canada (2):
  - McMaster University Medical Centre - Hamilton Health Sciences, Hamilton, Ontario
  - St. Michael's Hospital, Toronto, Ontario
- France (4):
  - CHRU de Brest - La Cavale Blanche, Brest
  - Hôpital Cardiologique Louis Pradel, Bron
  - CHU Hôtel-Dieu, Nantes
  - Hopital Necker, Hematologie Adultes, Paris
- Germany (4):
  - Vivantes Klinikum Friedrichshain, Berlin
  - Universitatsklinikum Bonn. Anstalt des oeffentlichen Rechts, Bonn
  - Universitaetsklinikum Giessen, Giessen
  - Universität und Universitätsklinikum des Saarlandes, Homburg/Saar
- Greece (2):
  - General Hospital of Athens "Hippokration", Athens, Attica
  - General Hospital of Athens "LAIKO", 2nd Regional Blood Transfusion Center, Athens, Attica
- The Chaim Sheba Medical Center, The National Hemophilia Center, Tel Litwinsky, Israel
- Italy (4):
  - IRCCS - AOU di Bologna, Policlinico di Sant'Orsola, Bologna, BO
  - UOC Medicina Interna - Malattie Emorragiche e Trombotiche, Napoli, Naples
  - SODc. Malattie Emorragiche e della Coagulazione Centro di Riferimento Regionale per le, Florence
  - Università degli studi di Roma "La Sapienza"- Policlinico Umberto I, Roma
- Japan (6):
  - Nagoya University Hospital - Transfusion Medicine, Nagoya, Aichi-ken
  - Sapporo Tokushukai Hospital, Sapporo, Hokkaido
  - Nara Medical University Hospital, Kashihara, Nara
  - Saitama Medical University Hospital, Iruma-gun, Saitama
  - National Center for Child Health and Development, Setagaya-ku, Tokyo
  - Ogikubo Hospital, Suginami-ku, Tokyo
- Saudi Arabia (2):
  - King Abdulaziz Medical City, Riyadh
  - King Faisal Specialist Hospital & Research Center, Riyadh
- South Korea (3):
  - Kyungpook National University Hospital, Daegu
  - Severance Hospital, Yonsei University Health System, Seoul
  - Kyung Hee University Hospital At Gangdong, Seoul
- Spain (5):
  - Hospital Universitario Virgen de la Arrixaca, El Palmar, Murcia
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari Vall d´Hebrón, Barcelona
  - H.U. La Paz., Madrid
  - H.U. Rio Hortega, Valladolid
- Skåne University Hospital, Malmo, Sweden
- Taiwan (5):
  - Changhua Christian Hospital, Changhua
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Chung Shan Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
- Turkey (Türkiye) (6):
  - Ege Universitesi Tip Fakultesi Cocuk Sagligi Ve Hastaliklari Anabilim Dali Pediatric Hematoloji, Bornova, İ̇zmir
  - Ege Universitesi Tip Fakultesi Hematoloji BD, Bornova, İ̇zmir
  - Acibadem Adana Hospital, Department of Pediatric Hematology, Adana
  - Akdeniz University Medical Faculty Hospital, Antalya
  - Gaziantep University Sahinbey Training and Research Hospital, Gaziantep
  - Istanbul University Oncology Institute, Istanbul
- United Kingdom (5):
  - Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne, TYNE & WEAR
  - Non Malignant Haematology Research Unit, Newcastle upon Tyne, TYNE & WEAR
  - Clinical Research Facility, Glasgow
  - Department of Haematology, Glasgow
  - Guy's and St Thomas' NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C0371004

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard of Care FIX Replacement Therapy (Hemophilia B): Participants with moderately severe to severe hemophilia B who administered their own current Factor IX (FIX) replacement therapy in the usual healthcare setting were included. No investigational product was administered as a part of this study.
- Standard of Care FVIII Replacement Therapy (Hemophilia A): Participants with moderately severe to severe hemophilia A who administered their own current Factor VIII (FVIII) replacement therapy in the usual healthcare setting were included. No investigational product was administered as a part of this study.
Period: Overall Study
Arm/Group | Standard of Care FIX Replacement Therapy (Hemophilia B) | Standard of Care FVIII Replacement Therapy (Hemophilia A)
Started | 111 | 101
Safety Analysis Set | 111 | 101
Efficacy Analysis Set | 110 | 96
Per-protocol Analysis Set | 107 | 81
Protocol Amendment 5 Analysis Set | 39 | 24
Completed | 107 | 99
Not Completed | 4 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — No Longer Met Eligibility Criteria | 0 | 1
Not completed — Withdrawal by Subject | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Standard of Care FIX Replacement Therapy (Hemophilia B): Participants with moderately severe to severe hemophilia B who administered their own current FIX replacement therapy in the usual healthcare setting were included. No investigational product was administered as a part of this study.
- Standard of Care FVIII Replacement Therapy (Hemophilia A): Participants with moderately severe to severe hemophilia A who administered their own current FVIII replacement therapy in the usual healthcare setting were included. No investigational product was administered as a part of this study.
- Total: Total of all reporting groups
Arm/Group | Standard of Care FIX Replacement Therapy (Hemophilia B) | Standard of Care FVIII Replacement Therapy (Hemophilia A) | Total
Number analyzed (Participants) | 111 | 101 | 212
Age, Customized [Count of Participants; unit: Participants]
  18-44 Years | 93 | 84 | 177
  45-64 Years | 18 | 17 | 35
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 111 | 101 | 212
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 8
  Not Hispanic or Latino | 91 | 76 | 167
  Unknown or Not Reported | 16 | 21 | 37
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 18 | 17 | 35
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 6 | 8
  White | 90 | 78 | 168
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Annualized Bleeding Rate (ABR) for Treated Bleeds and All Bleeds During Prospective Data Collection Period in Hemophilia B Participants: Efficacy Analysis Set
Description: ABR per participant was calculated as number of bleeds over number of days from baseline visit (Day 1 of the study) to end of study multiplication(*)365.25 days. All bleeds included treated and untreated bleeds. A treated bleed was defined as an event necessitating administration of coagulation factor within 72 hours of signs or symptoms of bleeding. An untreated bleed was defined as an event not necessitating administration of coagulation factor within 72 hours of signs or symptoms of bleeding. In this outcome measure, ABR for all and treated bleeds during prospective data collection period in hemophilia B participants per efficacy analysis set was reported. Abbreviations used: AAV6 = adeno-associated virus 6; AAV-Spark100 = Bioengineered AAV capsid, derived from a naturally occurring AAV serotype; nAb = neutralizing antibodies.
Time Frame: During prospective data collection period (from baseline visit of the study [Day 1] up to end of study follow-up [maximum follow-up: 1269 days])
Population: Efficacy analysis set: participants who signed an informed consent form (ICF), had their blood sample collected and assayed for AAV-Spark100 or AAV6 immunity testing, who were subsequently identified as nAb negative (negative for nAb to AAV-Spark100 for the hemophilia B cohort), met the inclusion/ exclusion criteria and who participated in the prospective data collection phase as part of their usual healthcare setting.
Measure: Mean (Standard Deviation); unit: Bleeds per year
Arm/Group | Standard of Care FIX Replacement Therapy (Hemophilia B)
Number analyzed (Participants) | 110
Bleeds per year
  Treated bleeds | 3.61 (7.634)
  All bleeds | 4.46 (9.446)

2. Primary Outcome: ABR for Treated Bleeds and All Bleeds During Prospective Data Collection Period in Hemophilia B Participants: Per-protocol Analysis Set
Description: ABR per participant was calculated as number of bleeds over number of days from baseline visit (Day 1 of the study) to end of study*365.25 days. All bleeds included treated and untreated bleeds. A treated bleed was defined as an event necessitating administration of coagulation factor within 72 hours of signs or symptoms of bleeding. An untreated bleed was defined as an event not necessitating administration of coagulation factor within 72 hours of signs or symptoms of bleeding. In this outcome measure, ABR for all and treated bleeds during prospective data collection period in hemophilia B participants per protocol analysis set was reported.
Time Frame: as for outcome 1
Population: Per-Protocol analysis set: all participants who signed an ICF, had their blood sample collected and assayed for AAV-Spark100 or AAV6 immunity testing, who were subsequently identified as nAb negative (negative for nAb to AAV-Spark100 for the hemophilia B cohort), met the inclusion/ exclusion criteria and who participated and completed at least 6 months of the prospective data collection phase as part of their usual healthcare setting.
Measure: Mean (Standard Deviation); unit: Bleeds per year
Arm/Group | Standard of Care FIX Replacement Therapy (Hemophilia B)
Number analyzed (Participants) | 107
Bleeds per year
  Treated bleeds | 3.71 (7.717)
  All bleeds | 4.56 (9.557)

3. Primary Outcome: ABR for Treated Bleeds and All Bleeds During Prospective Data Collection Period in Hemophilia B Participants: Protocol Amendment 5 Analysis Set
Description: ABR per participant was calculated as number of bleeds over number of days from baseline visit (Day 1 of the study) to end of study*365.25 days. All bleeds included treated and untreated bleeds. A treated bleed was defined as an event necessitating administration of coagulation factor within 72 hours of signs or symptoms of bleeding. An untreated bleed was defined as an event not necessitating administration of coagulation factor within 72 hours of signs or symptoms of bleeding. In this outcome measure, ABR for all and treated bleeds during prospective data collection period in hemophilia B participants per protocol amendment 5 analysis set was reported.
Time Frame: as for outcome 1
Population: Protocol Amendment 5 analysis set: all participants enrolled under Protocol Amendment 5 and afterwards, who fulfilled the inclusion/exclusion criteria and had prospective data collected.
Measure: Mean (Standard Deviation); unit: Bleeds per year
Arm/Group | Standard of Care FIX Replacement Therapy (Hemophilia B)
Number analyzed (Participants) | 39
Bleeds per year
  Treated bleeds | 4.21 (10.609)
  All bleeds | 4.78 (10.887)

4. Primary Outcome: ABR for Treated Bleeds and All Bleeds During Retrospective Data Collection Period in Hemophilia B Participants: Protocol Amendment 5 Analysis Set
Description: ABR per participant was calculated as number of bleeds over number of days from baseline visit (Day 1 of the study) to end of study*365.25 days. All bleeds included treated and untreated bleeds. A treated bleed was defined as an event necessitating administration of coagulation factor within 72 hours of signs or symptoms of bleeding. An untreated bleed was defined as an event not necessitating administration of coagulation factor within 72 hours of signs or symptoms of bleeding. In this outcome measure, ABR for all and treated bleeds during retrospective data collection period in hemophilia B participants per protocol amendment 5 analysis set was reported.
Time Frame: During retrospective data collection period (12 months before screening collected in the hemophilia history case report form [CRF])
Population: Protocol Amendment 5 analysis set: all participants enrolled under Protocol Amendment 5 and afterwards, who fulfilled the inclusion/exclusion criteria and had retrospective data collected. Here, "Overall Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Bleeds per year
Arm/Group | Standard of Care FIX Replacement Therapy (Hemophilia B)
Number analyzed (Participants) | 38
Bleeds per year
  Treated bleeds | 5.42 (8.163)
  All bleeds | 6.79 (10.390)

5. Primary Outcome: ABR for Treated Bleeds and All Bleeds From the Combined Retrospective and Prospective Data Collection Period in Hemophilia B Participants: Protocol Amendment 5 Analysis Set
Description: ABR per participant was calculated as number of bleeds over number of days from baseline visit (Day 1 of the study) to end of study*365.25 days. All bleeds included treated and untreated bleeds. A treated bleed was defined as an event necessitating administration of coagulation factor within 72 hours of signs or symptoms of bleeding. An untreated bleed was defined as an event not necessitating administration of coagulation factor within 72 hours of signs or symptoms of bleeding. In this outcome measure, ABR for all and treated bleeds during retrospective and prospective data collection period in hemophilia B participants per protocol amendment 5 analysis set was reported.
Time Frame: From start of retrospective data collection period (12 months before screening collected in hemophilia history CRF) up to end of prospective data collection follow-up of period (maximum follow-up:1269 days), for a total of approximately 4.5 years
Population: Protocol Amendment 5 analysis set: all participants enrolled under Protocol Amendment 5 and afterwards, who fulfilled the inclusion/exclusion criteria and had retrospective and prospective data collected. Here, "Overall Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Bleeds per year
Arm/Group | Standard of Care FIX Replacement Therapy (Hemophilia B)
Number analyzed (Participants) | 38
Bleeds per year
  Treated bleeds | 4.65 (7.589)
  All bleeds | 5.48 (8.284)

6. Primary Outcome: ABR for Treated Bleeds and All Bleeds During Prospective Data Collection Period in Hemophilia A Participants: Efficacy Analysis Set
Description: ABR per participant was calculated as number of bleeds over number of days from baseline visit (Day 1 of the study) to end of study*365.25 days. All bleeds included treated and untreated bleeds. A treated bleed was defined as an event necessitating administration of coagulation factor within 72 hours of signs or symptoms of bleeding. An untreated bleed was defined as an event not necessitating administration of coagulation factor within 72 hours of signs or symptoms of bleeding. In this outcome measure, ABR for all and treated bleeds during prospective data collection period in hemophilia A participants per efficacy analysis set was reported.
Time Frame: During prospective data collection period (from baseline visit of the study [Day 1] up to end of study follow-up [maximum follow-up: 948 days])
Population: Efficacy analysis set: participants who signed an ICF, had their blood sample collected and assayed for AAV-Spark100 or AAV6 immunity testing, who were subsequently identified as nAb negative (negative for nAb to AAV6 for the hemophilia A cohort), met the inclusion/ exclusion criteria and who participated in the prospective data collection phase as part of their usual healthcare setting.
Measure: Mean (Standard Deviation); unit: Bleeds per year
Arm/Group | Standard of Care FVIII Replacement Therapy (Hemophilia A)
Number analyzed (Participants) | 96
Bleeds per year
  Treated bleeds | 4.87 (7.246)
  All bleeds | 6.10 (10.578)

7. Primary Outcome: ABR for Treated Bleeds and All Bleeds During Prospective Data Collection Period in Hemophilia A Participants: Per-protocol Analysis Set
Description: ABR per participant was calculated as number of bleeds over number of days from baseline visit (Day 1 of the study) to end of study*365.25 days. All bleeds included treated and untreated bleeds. A treated bleed was defined as an event necessitating administration of coagulation factor within 72 hours of signs or symptoms of bleeding. An untreated bleed was defined as an event not necessitating administration of coagulation factor within 72 hours of signs or symptoms of bleeding. In this outcome measure, ABR for all and treated bleeds during prospective data collection period in hemophilia A participants per protocol analysis set was reported.
Time Frame: as for outcome 6
Population: Per-Protocol analysis set: all participants who signed an ICF, had their blood sample collected and assayed for AAV-Spark100 or AAV6 immunity testing, who were subsequently identified as nAb negative (negative for nAb to AAV6 for the hemophilia A cohort), met the inclusion/ exclusion criteria and who participated and completed at least 6 months of the prospective data collection phase as part of their usual healthcare setting.
Measure: Mean (Standard Deviation); unit: Bleeds per year
Arm/Group | Standard of Care FVIII Replacement Therapy (Hemophilia A)
Number analyzed (Participants) | 81
Bleeds per year
  Treated bleeds | 3.82 (5.665)
  All bleeds | 4.33 (6.700)

8. Primary Outcome: ABR for Treated Bleeds and All Bleeds During Prospective Data Collection Period in Hemophilia A Participants: Protocol Amendment 5 Analysis Set
Description: ABR per participant was calculated as number of bleeds over number of days from baseline visit (Day 1 of the study) to end of study*365.25 days. All bleeds included treated and untreated bleeds. A treated bleed was defined as an event necessitating administration of coagulation factor within 72 hours of signs or symptoms of bleeding. An untreated bleed was defined as an event not necessitating administration of coagulation factor within 72 hours of signs or symptoms of bleeding. In this outcome measure, ABR for all and treated bleeds during prospective data collection period in hemophilia A participants per protocol amendment 5 analysis set was reported.
Time Frame: as for outcome 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Bleeds per year
Arm/Group | Standard of Care FVIII Replacement Therapy (Hemophilia A)
Number analyzed (Participants) | 24
Bleeds per year
  Treated bleeds | 7.62 (9.907)
  All bleeds | 10.86 (16.692)

9. Primary Outcome: ABR for Treated Bleeds and All Bleeds During Retrospective Data Collection Period in Hemophilia A Participants: Protocol Amendment 5 Analysis Set
Description: ABR per participant was calculated as number of bleeds over number of days from baseline visit (Day 1 of the study) to end of study*365.25 days. All bleeds included treated and untreated bleeds. A treated bleed was defined as an event necessitating administration of coagulation factor within 72 hours of signs or symptoms of bleeding. An untreated bleed was defined as an event not necessitating administration of coagulation factor within 72 hours of signs or symptoms of bleeding. In this outcome measure, ABR for all and treated bleeds during retrospective data collection period in hemophilia A participants per protocol amendment 5 analysis set was reported.
Time Frame: During retrospective data collection period (12 months before screening collected in the hemophilia history CRF)
Population: Protocol Amendment 5 analysis set: all participants enrolled under Protocol Amendment 5 and afterwards, who fulfilled the inclusion/exclusion criteria and had retrospective data collected.
Measure: Mean (Standard Deviation); unit: Bleeds per year
Arm/Group | Standard of Care FVIII Replacement Therapy (Hemophilia A)
Number analyzed (Participants) | 24
Bleeds per year
  Treated bleeds | 9.83 (13.656)
  All bleeds | 14.29 (18.208)

10. Primary Outcome: ABR for Treated Bleeds and All Bleeds From the Combined Retrospective and Prospective Data Collection Period in Hemophilia A Participants: Protocol Amendment 5 Analysis Set
Description: ABR per participant was calculated as number of bleeds over number of days from baseline visit (Day 1 of the study) to end of study*365.25 days. All bleeds included treated and untreated bleeds. A treated bleed was defined as an event necessitating administration of coagulation factor within 72 hours of signs or symptoms of bleeding. An untreated bleed was defined as an event not necessitating administration of coagulation factor within 72 hours of signs or symptoms of bleeding. In this outcome measure, ABR for all and treated bleeds during retrospective and prospective data collection period in hemophilia A participants per protocol amendment 5 analysis set was reported.
Time Frame: From start of retrospective data collection period (12 months before screening collected in hemophilia history CRF) up to end of prospective data collection follow-up of period (maximum follow-up:948 days), for a total of approximately 3.6 years
Population: Protocol Amendment 5 analysis set: all participants enrolled under Protocol Amendment 5 and afterwards, who fulfilled the inclusion/exclusion criteria and had retrospective and prospective data collected.
Measure: Mean (Standard Deviation); unit: Bleeds per year
Arm/Group | Standard of Care FVIII Replacement Therapy (Hemophilia A)
Number analyzed (Participants) | 24
Bleeds per year
  Treated bleeds | 9.01 (11.908)
  All bleeds | 12.77 (16.290)

11. Secondary Outcome: Annualized Infusion Rate (AIR) During Prospective Data Collection Period in Hemophilia B Participants: Efficacy Analysis Set
Description: AIR per participant was calculated as the number of infusions received over number of days from baseline visit (Day 1) to end of study * 365.25 days.
Time Frame: as for outcome 1
Population: Efficacy analysis set: participants who signed an ICF, had their blood sample collected and assayed for AAV-Spark100 or AAV6 immunity testing, who were subsequently identified as nAb negative (negative for nAb to AAV-Spark100 for the hemophilia B cohort), met the inclusion/ exclusion criteria and who participated in the prospective data collection phase as part of their usual healthcare setting.
Measure: Mean (Standard Deviation); unit: Infusions per year
Arm/Group | Standard of Care FIX Replacement Therapy (Hemophilia B)
Number analyzed (Participants) | 110
Infusions per year | 62.81 (33.250)

12. Secondary Outcome: AIR During Prospective Data Collection Period in Hemophilia B Participants: Per-protocol Analysis Set
Description: as for outcome 11
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Infusions per year
Arm/Group | Standard of Care FIX Replacement Therapy (Hemophilia B)
Number analyzed (Participants) | 107
Infusions per year | 62.82 (33.213)

13. Secondary Outcome: AIR During Prospective Data Collection Period in Hemophilia B Participants: Protocol Amendment 5 Analysis Set
Description: as for outcome 11
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Infusions per year
Arm/Group | Standard of Care FIX Replacement Therapy (Hemophilia B)
Number analyzed (Participants) | 39
Infusions per year | 56.97 (20.987)

14. Secondary Outcome: AIR During Retrospective Data Collection Period in Hemophilia B Participants: Protocol Amendment 5 Analysis Set
Description: as for outcome 11
Time Frame: During retrospective data collection period (12 months before screening collected in the hemophilia history CRF)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Infusions per year
Arm/Group | Standard of Care FIX Replacement Therapy (Hemophilia B)
Number analyzed (Participants) | 39
Infusions per year | 66.97 (30.535)

15. Secondary Outcome: AIR From the Combined Retrospective and Prospective Data Collection Period in Hemophilia B Participants: Protocol Amendment 5 Analysis Set
Description: AIR combining retrospective and prospective data was calculated as (number of infusions from baseline visit (Day 1) to end of study + number of infusions collected in the Hemophilia History form) / (number of days from baseline visit (Day 1) to end of study + 365.25) / 365.25.
Time Frame: as for outcome 5
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Infusions per year
Arm/Group | Standard of Care FIX Replacement Therapy (Hemophilia B)
Number analyzed (Participants) | 39
Infusions per year | 60.98 (23.130)

16. Secondary Outcome: AIR During Prospective Data Collection Period in Hemophilia A Participants: Efficacy Analysis Set
Description: as for outcome 11
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Infusions per year
Arm/Group | Standard of Care FVIII Replacement Therapy (Hemophilia A)
Number analyzed (Participants) | 96
Infusions per year | 127.07 (51.784)

17. Secondary Outcome: AIR During Prospective Data Collection Period in Hemophilia A Participants: Per-protocol Analysis Set
Description: as for outcome 11
Time Frame: as for outcome 6
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Infusions per year
Arm/Group | Standard of Care FVIII Replacement Therapy (Hemophilia A)
Number analyzed (Participants) | 81
Infusions per year | 127.12 (55.418)

18. Secondary Outcome: AIR During Prospective Data Collection Period in Hemophilia A Participants: Protocol Amendment 5 Analysis Set
Description: as for outcome 11
Time Frame: as for outcome 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Infusions per year
Arm/Group | Standard of Care FVIII Replacement Therapy (Hemophilia A)
Number analyzed (Participants) | 24
Infusions per year | 133.19 (56.725)

19. Secondary Outcome: AIR During Retrospective Data Collection Period in Hemophilia A Participants: Protocol Amendment 5 Analysis Set
Description: as for outcome 11
Time Frame: During retrospective data collection period (12 months before screening collected in the hemophilia history CRF)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Infusions per year
Arm/Group | Standard of Care FVIII Replacement Therapy (Hemophilia A)
Number analyzed (Participants) | 24
Infusions per year | 141.88 (50.487)

20. Secondary Outcome: AIR From the Combined Retrospective and Prospective Data Collection Period in Hemophilia A Participants: Protocol Amendment 5 Analysis Set
Description: as for outcome 15
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Infusions per year
Arm/Group | Standard of Care FVIII Replacement Therapy (Hemophilia A)
Number analyzed (Participants) | 24
Infusions per year | 139.88 (52.490)

21. Secondary Outcome: Annualized Total Factor IX Replacement Therapy Consumption During Prospective Data Collection Period in Hemophilia B Participants: Efficacy Analysis Set
Description: Annualized factor consumption was calculated as the total factor replacement therapy consumption (in international unit [IU] and dose) *365.25 days/number of days during the observation time period while the participant received factor prophylaxis replacement therapy in the usual care setting from baseline visit (Day 1) to end of study.
Time Frame: as for outcome 1
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: International units per year
Arm/Group | Standard of Care FIX Replacement Therapy (Hemophilia B)
Number analyzed (Participants) | 110
International units per year | 238312 (127817)

22. Secondary Outcome: Annualized Total Factor IX Replacement Therapy Consumption During Prospective Data Collection Period in Hemophilia B Participants: Per-protocol Analysis Set
Description: Annualized factor consumption was calculated as the total factor replacement therapy consumption (in IU and dose) *365.25 days/number of days during the observation time period while the participant received factor prophylaxis replacement therapy in the usual care setting from baseline visit (Day 1) to end of study.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: International units per year
Arm/Group | Standard of Care FIX Replacement Therapy (Hemophilia B)
Number analyzed (Participants) | 107
International units per year | 240501 (128676)

23. Secondary Outcome: Annualized Total Factor IX Replacement Therapy Consumption During Prospective Data Collection Period in Hemophilia B Participants: Protocol Amendment 5 Analysis Set
Description: as for outcome 22
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: International units per year
Arm/Group | Standard of Care FIX Replacement Therapy (Hemophilia B)
Number analyzed (Participants) | 39
International units per year | 223408 (85995)

24. Secondary Outcome: Annualized Total Factor IX Replacement Therapy Consumption During Prospective Data Collection Period in Hemophilia A Participants: Efficacy Analysis Set
Description: as for outcome 22
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: International units per year
Arm/Group | Standard of Care FVIII Replacement Therapy (Hemophilia A)
Number analyzed (Participants) | 96
International units per year | 304998 (153932)

25. Secondary Outcome: Annualized Total Factor IX Replacement Therapy Consumption During Prospective Data Collection Period in Hemophilia A Participants: Per-protocol Analysis Set
Description: as for outcome 22
Time Frame: as for outcome 6
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: International units per year
Arm/Group | Standard of Care FVIII Replacement Therapy (Hemophilia A)
Number analyzed (Participants) | 81
International units per year | 314195 (163786)

26. Secondary Outcome: Annualized Total Factor IX Replacement Therapy Consumption During Prospective Data Collection Period in Hemophilia A Participants: Protocol Amendment 5 Analysis Set
Description: as for outcome 22
Time Frame: as for outcome 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: International units per year
Arm/Group | Standard of Care FVIII Replacement Therapy (Hemophilia A)
Number analyzed (Participants) | 24
International units per year | 235097 (67977)

27. Secondary Outcome: ABR for Spontaneous Treated Bleeds and All Bleeds During Prospective Data Collection Period in Hemophilia B Participants: Efficacy Analysis Set
Description: ABR per participant was calculated as number of bleeds over number of days from baseline visit (Day 1 of the study) to end of study*365.25 days. Spontaneous bleeds were defined as bleeding for no apparent or known reason particularly into the joints, muscles, and soft tissues. All bleeds included treated and untreated bleeds. A treated bleed was defined as an event necessitating administration of coagulation factor within 72 hours of signs or symptoms of bleeding. An untreated bleed was defined as an event not necessitating administration of coagulation factor within 72 hours of signs or symptoms of bleeding. In this outcome measure, ABR for spontaneous all and treated bleeds during prospective data collection period in hemophilia B participants per efficacy analysis set was reported.
Time Frame: as for outcome 1
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Bleeds per year
Arm/Group | Standard of Care FIX Replacement Therapy (Hemophilia B)
Number analyzed (Participants) | 110
Bleeds per year
  Treated bleeds | 2.11 (3.835)
  All bleeds | 2.79 (6.411)

28. Secondary Outcome: ABR for Traumatic Treated Bleeds and All Bleeds During Prospective Data Collection Period in Hemophilia B Participants: Efficacy Analysis Set
Description: ABR per participant was calculated as number of bleeds over number of days from baseline visit (Day 1 of the study) to end of study*365.25 days. Traumatic bleeds were defined as bleeding event occurring for an apparent or known reason. All bleeds included treated and untreated bleeds. A treated bleed was defined as an event necessitating administration of coagulation factor within 72 hours of signs or symptoms of bleeding. An untreated bleed was defined as an event not necessitating administration of coagulation factor within 72 hours of signs or symptoms of bleeding. In this outcome measure, ABR for traumatic all and treated bleeds during prospective data collection period in hemophilia B participants per efficacy analysis set was reported.
Time Frame: as for outcome 1
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Bleeds per year
Arm/Group | Standard of Care FIX Replacement Therapy (Hemophilia B)
Number analyzed (Participants) | 110
Bleeds per year
  Treated bleeds | 1.50 (6.380)
  All bleeds | 1.68 (6.623)

29. Secondary Outcome: ABR for Spontaneous Treated Bleeds and All Bleeds During Prospective Data Collection Period in Hemophilia B Participants: Per-protocol Analysis Set
Description: ABR per participant was calculated as number of bleeds over number of days from baseline visit (Day 1 of the study) to end of study*365.25 days. Spontaneous bleeds were defined as bleeding for no apparent or known reason particularly into the joints, muscles, and soft tissues. All bleeds included treated and untreated bleeds. A treated bleed was defined as an event necessitating administration of coagulation factor within 72 hours of signs or symptoms of bleeding. An untreated bleed was defined as an event not necessitating administration of coagulation factor within 72 hours of signs or symptoms of bleeding. In this outcome measure, ABR for spontaneous all and treated bleeds during prospective data collection period in hemophilia B participants per protocol analysis set was reported.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Bleeds per year
Arm/Group | Standard of Care FIX Replacement Therapy (Hemophilia B)
Number analyzed (Participants) | 107
Bleeds per year
  Treated bleeds | 2.17 (3.872)
  All bleeds | 2.84 (6.490)

30. Secondary Outcome: ABR for Traumatic Treated Bleeds and All Bleeds During Prospective Data Collection Period in Hemophilia B Participants: Per-protocol Analysis Set
Description: ABR per participant was calculated as number of bleeds over number of days from baseline visit (Day 1 of the study) to end of study*365.25 days. Traumatic bleeds were defined as bleeding event occurring for an apparent or known reason. All bleeds included treated and untreated bleeds. A treated bleed was defined as an event necessitating administration of coagulation factor within 72 hours of signs or symptoms of bleeding. An untreated bleed was defined as an event not necessitating administration of coagulation factor within 72 hours of signs or symptoms of bleeding. In this outcome measure, ABR for traumatic all and treated bleeds during prospective data collection period in hemophilia B participants per protocol analysis set was reported.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Bleeds per year
Arm/Group | Standard of Care FIX Replacement Therapy (Hemophilia B)
Number analyzed (Participants) | 107
Bleeds per year
  Treated bleeds | 1.54 (6.465)
  All bleeds | 1.72 (6.710)

31. Secondary Outcome: ABR for Spontaneous Treated Bleeds and All Bleeds During Prospective Data Collection Period in Hemophilia A Participants: Efficacy Analysis Set
Description: ABR per participant was calculated as number of bleeds over number of days from baseline visit (Day 1 of the study) to end of study*365.25 days. Spontaneous bleeds were defined as bleeding for no apparent or known reason particularly into the joints, muscles, and soft tissues. All bleeds included treated and untreated bleeds. A treated bleed was defined as an event necessitating administration of coagulation factor within 72 hours of signs or symptoms of bleeding. An untreated bleed was defined as an event not necessitating administration of coagulation factor within 72 hours of signs or symptoms of bleeding. In this outcome measure, ABR for spontaneous all and treated bleeds during prospective data collection period in hemophilia A participants per efficacy analysis set was reported.
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Bleeds per year
Arm/Group | Standard of Care FVIII Replacement Therapy (Hemophilia A)
Number analyzed (Participants) | 96
Bleeds per year
  Treated bleeds | 3.15 (5.948)
  All bleeds | 3.89 (7.552)

32. Secondary Outcome: ABR for Traumatic Treated Bleeds and All Bleeds During Prospective Data Collection Period in Hemophilia A Participants: Efficacy Analysis Set
Description: ABR per participant was calculated as number of bleeds over number of days from baseline visit (Day 1 of the study) to end of study*365.25 days. Traumatic bleeds were defined as bleeding event occurring for an apparent or known reason. All bleeds included treated and untreated bleeds. A treated bleed was defined as an event necessitating administration of coagulation factor within 72 hours of signs or symptoms of bleeding. An untreated bleed was defined as an event not necessitating administration of coagulation factor within 72 hours of signs or symptoms of bleeding. In this outcome measure, ABR for traumatic all and treated bleeds during prospective data collection period in hemophilia A participants per efficacy analysis set was reported.
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Bleeds per year
Arm/Group | Standard of Care FVIII Replacement Therapy (Hemophilia A)
Number analyzed (Participants) | 96
Bleeds per year
  Treated bleeds | 1.78 (3.893)
  All bleeds | 2.27 (5.503)

33. Secondary Outcome: ABR for Spontaneous Treated Bleeds and All Bleeds During Prospective Data Collection Period in Hemophilia A Participants: Per-protocol Analysis Set
Description: ABR per participant was calculated as number of bleeds over number of days from baseline visit (Day 1 of the study) to end of study*365.25 days. Spontaneous bleeds were defined as bleeding for no apparent or known reason particularly into the joints, muscles, and soft tissues. All bleeds included treated and untreated bleeds. A treated bleed was defined as an event necessitating administration of coagulation factor within 72 hours of signs or symptoms of bleeding. An untreated bleed was defined as an event not necessitating administration of coagulation factor within 72 hours of signs or symptoms of bleeding. In this outcome measure, ABR for spontaneous all and treated bleeds during prospective data collection period in hemophilia A participants per protocol analysis set was reported.
Time Frame: as for outcome 6
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Bleeds per year
Arm/Group | Standard of Care FVIII Replacement Therapy (Hemophilia A)
Number analyzed (Participants) | 81
Bleeds per year
  Treated bleeds | 2.37 (4.101)
  All bleeds | 2.73 (5.143)

34. Secondary Outcome: ABR for Traumatic Treated Bleeds and All Bleeds During Prospective Data Collection Period in Hemophilia A Participants: Per-protocol Analysis Set
Description: ABR per participant was calculated as number of bleeds over number of days from baseline visit (Day 1 of the study) to end of study*365.25 days. Traumatic bleeds were defined as bleeding event occurring for an apparent or known reason. All bleeds included treated and untreated bleeds. A treated bleed was defined as an event necessitating administration of coagulation factor within 72 hours of signs or symptoms of bleeding. An untreated bleed was defined as an event not necessitating administration of coagulation factor within 72 hours of signs or symptoms of bleeding. In this outcome measure, ABR for traumatic all and treated bleeds during prospective data collection period in hemophilia A participants per protocol analysis set was reported.
Time Frame: as for outcome 6
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Bleeds per year
Arm/Group | Standard of Care FVIII Replacement Therapy (Hemophilia A)
Number analyzed (Participants) | 81
Bleeds per year
  Treated bleeds | 1.45 (3.467)
  All bleeds | 1.60 (3.608)

35. Other Pre Specified Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a study participant administered a product or medical device; the event need not necessarily have a causal relationship with the treatment or usage. An SAE was any untoward medical occurrence at any dose that met 1 of the following criteria: resulted in death; was life-threatening; required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/ incapacity; resulted in congenital anomaly/birth defect; other important medical events per protocol of the study.
Time Frame: During prospective data collection period: Day 1 through end of study visit (from baseline visit of the study [Day 1] up to end of study follow-up [maximum follow-up: 1269 days])
Population: Safety analysis set included all enrolled participants (negative for nAb to AAV-Spark100 for the hemophilia B cohort, or negative for nAb to AAV6 for the hemophilia A cohort) who entered the prospective data collection phase.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care FIX Replacement Therapy (Hemophilia B) | Standard of Care FVIII Replacement Therapy (Hemophilia A)
Number analyzed (Participants) | 111 | 101
Participants | 9 | 4

36. Other Pre Specified Outcome: Number of Participants With Adverse Events of Special Interest (AESIs)
Description: An AE was any untoward medical occurrence in a study participant administered a product or medical device; the event need not necessarily have a causal relationship with the treatment or usage. Adverse events of special interest are FIX/FVIII inhibitor development, thrombotic events, and FIX hypersensitivity events for this study.
Time Frame: as for outcome 35
Population: as for outcome 35
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care FIX Replacement Therapy (Hemophilia B) | Standard of Care FVIII Replacement Therapy (Hemophilia A)
Number analyzed (Participants) | 111 | 101
Participants | 2 | 0

ADVERSE EVENTS:
Time Frame: During prospective data collection period (from baseline visit of the study [Day 1] up to end of study follow-up [maximum follow-up: 1269 days])
Description: Same event may occur as both non-SAE and SAE but are distinct events. An event may be categorised as serious in 1 participant and non-serious in another, or a participant may have experienced both SAE and non-SAE. Safety analysis set was evaluated.
Arm/Group | Standard of Care FIX Replacement Therapy (Hemophilia B) | Standard of Care FVIII Replacement Therapy (Hemophilia A)
All-Cause Mortality (participants affected / at risk) | 0/111 | 0/101
Serious Adverse Events (participants affected / at risk) | 9/111 | 4/101
Other Adverse Events (participants affected / at risk) | 4/111 | 0/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard of Care FIX Replacement Therapy (Hemophilia B) (N=111) | Standard of Care FVIII Replacement Therapy (Hemophilia A) (N=101)
Enteritis (Gastrointestinal disorders) | 1 | 0 — MedDRA v27.1 was used for Hemophilia B cohort. MedDRA v26.0 was used for Hemophilia A cohort.
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0 — MedDRA v27.1 was used for Hemophilia B cohort. MedDRA v26.0 was used for Hemophilia A cohort.
Appendicitis (Infections and infestations) | 1 | 0 — MedDRA v27.1 was used for Hemophilia B cohort. MedDRA v26.0 was used for Hemophilia A cohort.
Joint injury (Injury, poisoning and procedural complications) | 1 | 0 — MedDRA v27.1 was used for Hemophilia B cohort. MedDRA v26.0 was used for Hemophilia A cohort.
Ligament rupture (Injury, poisoning and procedural complications) | 1 | 0 — MedDRA v27.1 was used for Hemophilia B cohort. MedDRA v26.0 was used for Hemophilia A cohort.
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 — MedDRA v27.1 was used for Hemophilia B cohort. MedDRA v26.0 was used for Hemophilia A cohort.
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 0 — MedDRA v27.1 was used for Hemophilia B cohort. MedDRA v26.0 was used for Hemophilia A cohort.
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 — MedDRA v27.1 was used for Hemophilia B cohort. MedDRA v26.0 was used for Hemophilia A cohort.
Haemophilic arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 — MedDRA v27.1 was used for Hemophilia B cohort. MedDRA v26.0 was used for Hemophilia A cohort.
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — MedDRA v27.1 was used for Hemophilia B cohort. MedDRA v26.0 was used for Hemophilia A cohort.
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1 — MedDRA v27.1 was used for Hemophilia B cohort. MedDRA v26.0 was used for Hemophilia A cohort.
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 — MedDRA v27.1 was used for Hemophilia B cohort. MedDRA v26.0 was used for Hemophilia A cohort.
Wound infection (Infections and infestations) | 0 | 1 — MedDRA v27.1 was used for Hemophilia B cohort. MedDRA v26.0 was used for Hemophilia A cohort.
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 — MedDRA v27.1 was used for Hemophilia B cohort. MedDRA v26.0 was used for Hemophilia A cohort.
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Standard of Care FIX Replacement Therapy (Hemophilia B) (N=111) | Standard of Care FVIII Replacement Therapy (Hemophilia A) (N=101)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 — MedDRA v27.1 was used for Hemophilia B cohort. MedDRA v26.0 was used for Hemophilia A cohort.
Haematoma (Vascular disorders) | 2 | 0 — MedDRA v27.1 was used for Hemophilia B cohort. MedDRA v26.0 was used for Hemophilia A cohort.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2023-03-31): https://cdn.clinicaltrials.gov/large-docs/16/NCT03587116/Prot_000.pdf
  • Statistical Analysis Plan (2024-09-19): https://cdn.clinicaltrials.gov/large-docs/16/NCT03587116/SAP_001.pdf